CLINICAL TRIAL: NCT02455310
Title: Extension Connection: Dissemination Effectiveness Evaluation
Brief Title: Extension Connection Evaluation
Acronym: ExConEval
Status: Completed | Type: Observational
Sponsor: Ryan M. Carnahan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Iowa State University (Other)
Responsible Party: Sponsor-Investigator, Ryan M. Carnahan, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201108751
Record Dates: First submitted 2015-04-30; First posted 2015-05-27 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Outpatients with dementia: Medication use will be evaluated among outpatients with dementia in intervention and control counties, as well as statewide to evaluate the long-term effectiveness of the statewide intervention.
  Interventions: Behavioral: Educational activities to improve dementia care
- Nursing home residents: Medication use and behavioral outcomes will be evaluated among nursing home residents in intervention and control counties, as well as statewide to evaluate the long-term effectiveness of the statewide intervention.
  Interventions: Behavioral: Educational activities to improve dementia care

INTERVENTIONS:
Behavioral: Educational activities to improve dementia care — The multicomponent intervention included active dissemination of educational resources and optional participation in specialist consultation sessions for up to 6 months. The standard intervention included education through a website or conferences, including clinical tools to support implementation of best practices.

SUMMARY:
This study will perform a retrospective analysis to evaluate the effectiveness of a multicomponent educational intervention to improve medication use and management of behavioral and psychological symptoms of dementia, relative to a statewide intervention that has been ongoing. Medication use and symptom severity outcomes will be compared among intervention counties and demographically similar non-intervention counties.

DETAILED DESCRIPTION:
This study will perform a retrospective analysis to evaluate the effectiveness of a multicomponent educational intervention to improve medication use and management of behavioral and psychological symptoms of dementia, relative to a statewide intervention that has been ongoing. Medication use and symptom severity outcomes will be compared among 29 intervention counties and 10 demographically similar non-intervention counties. The long-term effectiveness of the statewide intervention will also be evaluated. Medicare and Minimum Data set data from 2011 to 2014 will be used to evaluate prescribing and other outcomes in 1) outpatients with dementia, and 2) nursing home residents, based on exposure to interventions among healthcare and nursing home providers. Measurable goals included increasing the appropriateness of antipsychotic prescribing and reducing anticholinergic use. Effect modification will be evaluated by level of participation in the intervention and other prescriber and nursing home facility characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Current Medicare fee-for-service plan and Part D enrollment for at least 3 months prior to the month of interest and during the month of interest (allowing a gap of one month to be considered as continuous enrollment if the person is enrolled during the month of interest)
2. Age greater than or equal to 66 years at the end of a year of interest
3. Any dementia diagnosis prior to the month of interest, or current resident of a nursing home
4. For the nursing home analysis, at least 14 days in the facility in the month being classified

Exclusion Criteria:

1. Greater than 15 days of the month of interest when prescription fills are unobservable from Medicare Part D claims due to hospital inpatient status, skilled nursing facility resident status, or hospice enrollment
2. A diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, Huntington's disease, Down's syndrome, or mental retardation or developmental disability at any time during the study period. Diagnoses after entry into the study sample will be included because of the limited look-back period to define some conditions for some individuals, and because these are generally not conditions with late-life onset so they are assumed to have been present prior to the first occurrence of a diagnosis in the available data
3. Currently comatose based on the most recent MDS assessment-if currently in a nursing home

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All Iowa Medicare beneficiaries who are nursing home residents or diagnosed with dementia and meet other eligibility criteria, for each year from 2011 to 2014.
Sampling Method: Non-Probability Sample
Enrollment: 44524 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Antipsychotic use | Up to 4 years
  Antipsychotic use
Anticholinergic Use | Up to 4 years
  Anticholinergic use

SECONDARY OUTCOMES:
Olanzapine use in patients with metabolic disorders | Up to 4 years
  Proportion of antipsychotic users with diabetes mellitus, hyperlipidemia, or hypertension (based on diagnosis indicators from claims) who receive olanzapine, the least appropriate antipsychotic when these conditions are present due to its metabolic effects.
Excessive antipsychotic dose | Up to 4 years
  Antipsychotic doses as defined as excessive by CMS standards for nursing home residents with dementia
Benzodiazepine use | Up to 2 years
  Benzodiazepine use. Time frame differs because Medicare Part D did not pay for these drugs until 2013.
Quetiapine or clozapine use only among antipsychotic users with Parkinson's disease or Lewy body dementia | Up to 4 years
  Quetiapine or clozapine use only among antipsychotic users with Parkinson's disease or Lewy body dementia. These are the most appropriate antipsychotics in these conditions.
Antipsychotic use in people with dementia | Up to 4 years
  Antipsychotic use in people with dementia. This is a subgroup analysis of the nursing home population.
Antipsychotic use in nursing home residents with a potentially appropriate indication | Up to 4 years
  Proportion of antipsychotic users with evidence of a potentially appropriate indication, stratified by indication, as follows: verbal or physical aggression, delusions, hallucinations, delirium
Antipsychotic use in nursing home residents without a potentially appropriate indication, and proportion with evidence of an inappropriate indication | Up to 4 years
  Antipsychotic use in those without a potentially appropriate indication, and proportion of those users with evidence of an inappropriate indication
Antipsychotic use in nursing home residents with a recent history of falls | Up to 4 years
  Antipsychotic use in those with a recent history of falls (fall indicator on any MDS assessment in the prior 6 months)
Antipsychotic use in nursing home residents with an unsteady gait | Up to 4 years
  Antipsychotic use in nursing home residents with an unsteady gait, as evaluated by MDS records
Hypnotic use | Up to 4 years
  Hypnotic use as measured by MDS indicator
Changes in behavioral and psychological symptom presence | Up to 4 years
  Changes in behavioral symptom frequency (each of verbal aggression, physical aggression, delirium, hallucinations, delusions)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Carnahan, PharmD, MS, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa College of Public Health, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Other than exposure data which is identifiable, the evaluation is based on CMS data which cannot be shared without a data reuse agreement.